CLINICAL TRIAL: NCT02232282
Title: Acupuncture for Female Interstitial Cystitis/Painful Bladder Syndrome and Its Effect on the Urinary Microbiome: A Randomized Controlled Trial
Brief Title: Acupuncture for Female IC/PBSyndrome and Its Effect on the Urinary Microbiome: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Interstitial Cystitis Association (ICA) (Other)
Responsible Party: Principal Investigator, Larissa Bresler, M.D., Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206129
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Results first posted 2021-03-25 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis
Keywords: Painful Bladder Syndrome; Interstitial Cystitis; Suprapubic Pain; Urinary Urgency
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimal Acupuncture (Sham Comparator): Fifteen (15) will be allocated in the control sham/minimal acupuncture + standard medical treatments of IC. The sham intervention (also described as minimal intervention) will use superficial needle insertion at body locations not recognized as true acupoints. Patients will be explained that various acupuncture treatment protocols will be tested including "minimal acupuncture", therefore, the control group will not be aware of receiving sham acupuncture.
  Interventions: Device: Control Sham/Minimal Acupuncture
- Standard acupuncture treatment (Active Comparator): Fifteen (15) will be allocated in the standard acupuncture treatment + medical management of IC. Standard acupuncture treatment protocol will include 4 gates plus GV 20 to reduce anxiety and help with relaxation and to assess acupuncture naïve patient's response to needles during their first acupuncture encounter. Subsequent visits would include administration of curious meridian Chong Mo paired with Yang Ming. 4 Hz low level electrical stimulation will be applied.
  Interventions: Device: standard acupuncture treatment

INTERVENTIONS:
Device: standard acupuncture treatment — A standardized acupuncture treatment will be assigned, and both groups will receive 7 acupuncture treatments that follow a standardized protocol on classical acupuncture points, with or without mild electrical stimulation versus sham/minimal acupuncture. Acupuncture needles are single use, sterile and disposable. Standard acupuncture treatment protocol will include 4 gates plus GV 20 to reduce anxiety and help with relaxation and to assess acupuncture naïve patient's response to needles during their first acupuncture encounter. Subsequent visits would include administration of curious meridian Chong Mo paired with Yang Ming. 4 Hz low level electrical stimulation will be applied.
  Arms: Standard acupuncture treatment
Device: Control Sham/Minimal Acupuncture — Control group will receive sham/minimal acupuncture with low level electrical stimulation. The sham intervention (also described as minimal intervention) will use superficial needle insertion at body locations not recognized as true acupoints. Patients will be explained that various acupuncture treatment protocols will be tested including "minimal acupuncture", therefore, the control group will not be aware of receiving sham acupuncture. These described acupuncture treatments are well accepted treatment protocols for women with pelvic pain and bladder complaints.
  Arms: Minimal Acupuncture

SUMMARY:
The investigators central hypothesis is that women with Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS) will benefit from acupuncture compared with sham treatment and acupuncture responders will have a differential urinary microbiome.

DETAILED DESCRIPTION:
The Urinary Microbiota. Within internal surfaces, which are defined as existing outside the body (e.g. the intestinal epithelium or the vaginal epithelium), there exist commensal microbial communities. These microbiota are believed to be beneficial to human health, facilitating efficient removal of improperly functioning immune cells and protecting the host from pathogen infection13-15. The human bladder is a core component of the human urinary tract. It is a hollow muscular organ lined with transitional epithelium, which functions as the storage site for metabolic wastes in the form of urine. Given that the bladder's luminal space is also considered outside the body, it would seem reasonable that a urinary microbiota would be present. Yet, the historic dogma has maintained that urine is "sterile," based on culture-dependent methods of bacterial detection. This paradigm is shifting, however, based on our newly published data noting the presence of a urinary microbiota in adult women without clinical urinary tract infections16,17. Furthermore, we have recently discovered that the microbiota of women with overactive bladder (specifically with associated urgency incontinence) is distinguishable from the microbiota of women with stress urinary incontinence. These findings suggest that IC/PBS may be influenced by an alteration to the urinary microbiota. Indeed, recent evidence reports a difference in the urinary microbiome dominated by Lactobacillus in subjects with IC/PBS compared with healthy controls18. This work is limited by lack of correlative clinical symptomatology, small sample size and urinary samples that may have been contaminated.

The investigators long term goal is to determine pelvic pain mechanisms that will inform clinically-relevant classification and evidence-based treatment of women with IC/PBS and CPP. The short term goal of this application is to determine the safety, tolerability and efficacy of acupuncture in women with IC/PBS as a neuromodulative treatment and to correlate the urinary microbiome with acupuncture responders. Our approach will advance the understanding of the contribution and consequences of peripheral pelvic nociception in IC/PBS.

ELIGIBILITY:
Inclusion Criteria:

* Females, age 21 to 65 years
* Symptoms of urinary frequency, urgency and suprapubic/bladder pain for > 6 months
* Generally stable health
* An average bladder pain score of at least >3/10

Exclusion Criteria:

* Patients with pacemaker or other neurostimulator (gastric/spinal)
* History or current symptomatic urethral stricture, cystitis caused by tuberculosis, radiation therapy or Cytoxan/cyclophosphamide therapy
* Prior augmentation cystoplasty or cystectomy
* Systemic autoimmune disorder (such as Crohn's Disease, Ulcerative Colitis, Lupus, Rheumatoid Arthritis, or Multiple Sclerosis)
* Systemic neuromuscular disease known to affect the lower urinary tract
* History of urogenital cancer (with the exception of minor skin cancer)
* Current or imminent planned pregnancy/recent delivery <6 months
* Current pelvic floor physical therapy
* Current use of opioid medications (short or long acting) for pain
* Abdominal or pelvic surgery within the last 6 months.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Bresler, MD, Principal Investigator — Loyola University Medical Center Dept of Urology
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogart LM, Berry SH, Clemens JQ. Symptoms of interstitial cystitis, painful bladder syndrome and similar diseases in women: a systematic review. J Urol. 2007 Feb;177(2):450-6. doi: 10.1016/j.juro.2006.09.032. PMID 17222607
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Suskind AM, Berry SH, Suttorp MJ, Elliott MN, Hays RD, Ewing BA, Clemens JQ. Health-related quality of life in patients with interstitial cystitis/bladder pain syndrome and frequently associated comorbidities. Qual Life Res. 2013 Sep;22(7):1537-41. doi: 10.1007/s11136-012-0285-5. Epub 2012 Oct 7. PMID 23054497
- [Background] Adams K, Denman MA. Bladder pain syndrome: a review. Female Pelvic Med Reconstr Surg. 2011 Nov;17(6):279-89. doi: 10.1097/SPV.0b013e31823a8174. PMID 22453222
- [Background] Lai HH, North CS, Andriole GL, Sayuk GS, Hong BA. Polysymptomatic, polysyndromic presentation of patients with urological chronic pelvic pain syndrome. J Urol. 2012 Jun;187(6):2106-12. doi: 10.1016/j.juro.2012.01.081. Epub 2012 Apr 12. PMID 22503014
- [Background] Hoffman D. Understanding multisymptom presentations in chronic pelvic pain: the inter-relationships between the viscera and myofascial pelvic floor dysfunction. Curr Pain Headache Rep. 2011 Oct;15(5):343-6. doi: 10.1007/s11916-011-0215-1. PMID 21739128
- [Background] Warren JW, van de Merwe JP, Nickel JC. Interstitial cystitis/bladder pain syndrome and nonbladder syndromes: facts and hypotheses. Urology. 2011 Oct;78(4):727-32. doi: 10.1016/j.urology.2011.06.014. No abstract available. PMID 21855966
- [Background] Birder L, de Groat W, Mills I, Morrison J, Thor K, Drake M. Neural control of the lower urinary tract: peripheral and spinal mechanisms. Neurourol Urodyn. 2010;29(1):128-39. doi: 10.1002/nau.20837. PMID 20025024
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] O'Hare PG 3rd, Hoffmann AR, Allen P, Gordon B, Salin L, Whitmore K. Interstitial cystitis patients' use and rating of complementary and alternative medicine therapies. Int Urogynecol J. 2013 Jun;24(6):977-82. doi: 10.1007/s00192-012-1966-x. Epub 2012 Nov 14. PMID 23149598
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186
- [Background] Capodice JL, Jin Z, Bemis DL, Samadi D, Stone BA, Kapan S, Katz AE. A pilot study on acupuncture for lower urinary tract symptoms related to chronic prostatitis/chronic pelvic pain. Chin Med. 2007 Feb 6;2:1. doi: 10.1186/1749-8546-2-1. PMID 17284322
- [Background] Flint HJ, Scott KP, Louis P, Duncan SH. The role of the gut microbiota in nutrition and health. Nat Rev Gastroenterol Hepatol. 2012 Sep 4;9(10):577-89. doi: 10.1038/nrgastro.2012.156. eCollection 2012 Oct. PMID 22945443
- [Background] Frank DN, Zhu W, Sartor RB, Li E. Investigating the biological and clinical significance of human dysbioses. Trends Microbiol. 2011 Sep;19(9):427-34. doi: 10.1016/j.tim.2011.06.005. Epub 2011 Jul 19. PMID 21775143
- [Background] Gajer P, Brotman RM, Bai G, Sakamoto J, Schutte UM, Zhong X, Koenig SS, Fu L, Ma ZS, Zhou X, Abdo Z, Forney LJ, Ravel J. Temporal dynamics of the human vaginal microbiota. Sci Transl Med. 2012 May 2;4(132):132ra52. doi: 10.1126/scitranslmed.3003605. PMID 22553250
- [Background] Wolfe AJ, Toh E, Shibata N, Rong R, Kenton K, Fitzgerald M, Mueller ER, Schreckenberger P, Dong Q, Nelson DE, Brubaker L. Evidence of uncultivated bacteria in the adult female bladder. J Clin Microbiol. 2012 Apr;50(4):1376-83. doi: 10.1128/JCM.05852-11. Epub 2012 Jan 25. PMID 22278835
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Siddiqui H, Lagesen K, Nederbragt AJ, Jeansson SL, Jakobsen KS. Alterations of microbiota in urine from women with interstitial cystitis. BMC Microbiol. 2012 Sep 13;12:205. doi: 10.1186/1471-2180-12-205. PMID 22974186
- [Background] Zhang R, Lao L, Ren K, Berman BM. Mechanisms of acupuncture-electroacupuncture on persistent pain. Anesthesiology. 2014 Feb;120(2):482-503. doi: 10.1097/ALN.0000000000000101. PMID 24322588
- [Background] Kim SK, Bae H. Acupuncture and immune modulation. Auton Neurosci. 2010 Oct 28;157(1-2):38-41. doi: 10.1016/j.autneu.2010.03.010. Epub 2010 Apr 15. PMID 20399151
- [Background] Tyagi P, Killinger K, Tyagi V, Nirmal J, Chancellor M, Peters KM. Urinary chemokines as noninvasive predictors of ulcerative interstitial cystitis. J Urol. 2012 Jun;187(6):2243-8. doi: 10.1016/j.juro.2012.01.034. Epub 2012 Apr 13. PMID 22503040
- [Background] Lamale LM, Lutgendorf SK, Zimmerman MB, Kreder KJ. Interleukin-6, histamine, and methylhistamine as diagnostic markers for interstitial cystitis. Urology. 2006 Oct;68(4):702-6. doi: 10.1016/j.urology.2006.04.033. PMID 17070335
- [Background] Masters Steedman S, Middaugh SJ, Kee WG, Carson DS, Harden RN, Miller MC. Chronic-pain medications: equivalence levels and method of quantifying usage. Clin J Pain. 1992 Sep;8(3):204-14. PMID 1421733
- [Background] Gallizzi M, Gagnon C, Harden RN, Stanos S, Khan A. Medication Quantification Scale Version III: internal validation of detriment weights using a chronic pain population. Pain Pract. 2008 Jan-Feb;8(1):1-4. doi: 10.1111/j.1533-2500.2007.00163.x. PMID 18211588
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Huskisson EC. Measurement of pain. J Rheumatol. 1982 Sep-Oct;9(5):768-9. No abstract available. PMID 6184474
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Jerome A, Gross RT. Pain disability index: construct and discriminant validity. Arch Phys Med Rehabil. 1991 Oct;72(11):920-2. doi: 10.1016/0003-9993(91)90012-8. PMID 1929812
- [Background] FitzGerald MP, Anderson RU, Potts J, Payne CK, Peters KM, Clemens JQ, Kotarinos R, Fraser L, Cosby A, Fortman C, Neville C, Badillo S, Odabachian L, Sanfield A, O'Dougherty B, Halle-Podell R, Cen L, Chuai S, Landis JR, Mickelberg K, Barrell T, Kusek JW, Nyberg LM; Urological Pelvic Pain Collaborative Research Network. Randomized multicenter feasibility trial of myofascial physical therapy for the treatment of urological chronic pelvic pain syndromes. J Urol. 2009 Aug;182(2):570-80. doi: 10.1016/j.juro.2009.04.022. Epub 2009 Jun 17. PMID 19535099
- [Background] Clemens JQ, Calhoun EA, Litwin MS, McNaughton-Collins M, Kusek JW, Crowley EM, Landis JR; Urologic Pelvic Pain Collaborative Research Network. Validation of a modified National Institutes of Health chronic prostatitis symptom index to assess genitourinary pain in both men and women. Urology. 2009 Nov;74(5):983-7, quiz 987.e1-3. doi: 10.1016/j.urology.2009.06.078. Epub 2009 Oct 2. PMID 19800663
- [Background] O'Leary MP, Sant GR, Fowler FJ Jr, Whitmore KE, Spolarich-Kroll J. The interstitial cystitis symptom index and problem index. Urology. 1997 May;49(5A Suppl):58-63. doi: 10.1016/s0090-4295(99)80333-1. PMID 9146003
- [Background] Rosen RC. Measurement of male and female sexual dysfunction. Curr Psychiatry Rep. 2001 Jun;3(3):182-7. doi: 10.1007/s11920-001-0050-x. PMID 11353580
- [Background] Sullivan MJ, D'Eon JL. Relation between catastrophizing and depression in chronic pain patients. J Abnorm Psychol. 1990 Aug;99(3):260-3. doi: 10.1037//0021-843x.99.3.260. PMID 2145334
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Crew KD, Capodice JL, Greenlee H, Brafman L, Fuentes D, Awad D, Yann Tsai W, Hershman DL. Randomized, blinded, sham-controlled trial of acupuncture for the management of aromatase inhibitor-associated joint symptoms in women with early-stage breast cancer. J Clin Oncol. 2010 Mar 1;28(7):1154-60. doi: 10.1200/JCO.2009.23.4708. Epub 2010 Jan 25. PMID 20100963
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728

RESULTS

PARTICIPANT FLOW:
Groups:
- Minimal Acupuncture: This arm received sham/minimal acupuncture with low level electrical stimulation. This intervention used superficial needle insertion at body locations not recognized as true acupoints.
- Standard Acupuncture Treatment: This arm received standard acupuncture treatment: A standardized acupuncture treatment followed a standardized protocol on classical acupuncture points, with or without mild electrical stimulation Standard acupuncture treatment protocol will include 4 gates plus GV 20. Subsequent visits included administration of curious meridian Chong Mo paired with Yang Ming. 4 Hz low level electrical stimulation was applied.
Period: Overall Study
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment
Started | 10 | 12
Completed | 10 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (14.7) | 50.6 (12.1) | 49.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 6 | 9 | 15
  Race/Ethnicity: Hispanic | 2 | 1 | 3
  Race/Ethnicity: Black or African American | 1 | 0 | 1
  Race/Ethnicity: Other | 1 | 0 | 1
  Race/Ethnicity: Prefers not to answer | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Marital status [Count of Participants; unit: Participants]
  Married | 7 | 7 | 14
  Not married | 3 | 4 | 7
Education [Count of Participants; unit: Participants]
  Completed 4 years of college or more | 8 | 6 | 14
  Completed fewer than 4 years of college | 2 | 5 | 7
Body mass index [Median (Full Range); unit: kg/m^2] | 26.2 [19.1 to 38.0] | 24.0 [15.7 to 37.9] | 25.0 [15.7 to 38.0]
Menstrual status [Count of Participants; unit: Participants]
  Pre-menopausal | 5 | 5 | 10
  Post-menopausal | 5 | 5 | 10
  Not sure | 0 | 1 | 1
Vaginal parity [Count of Participants; unit: Participants]
  Nulliparous | 5 | 3 | 8
  At least primiparous | 5 | 8 | 13
Number of Pain comorbidities [Count of Participants; unit: Participants] — Pain comorbidities assessed include fibromyalgia, endometriosis, low back pain, vulvodynia, and irritable bowels
  Participants
    0 | 3 | 1 | 4
    1 | 3 | 3 | 6
    2 | 2 | 4 | 6
    3 | 2 | 2 | 4
    4 | 0 | 1 | 1
First line treatment [Count of Participants; unit: Participants] — Relaxation technique, yoga, diet
  Participants
    First-line treatment | 7 | 8 | 15
    No first-line treatment | 3 | 3 | 6
Second-line treatment [Count of Participants; unit: Participants] — pelvic floor physical therapy, biofeedback, amitriptyline, elimiron, bladder installation
  Participants
    Second-line treatment | 10 | 10 | 20
    No second-line treatment | 0 | 1 | 1
Third-line treatment [Count of Participants; unit: Participants] — hydrodistension
  Participants
    Third-line treatment | 5 | 5 | 10
    No third-line treatment | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Acupuncture to Reduce Pain in Women With Interstitial Cystitis/Painful Bladder Syndrome
Description: Change in worst pain as measured by the Brief Pain Inventory-Short Form. Scores range from 0 to 10 and higher scores indicate more pain. Change is calculated as the 6 weeks score minus the baseline score.
Time Frame: 0 weeks, 6 weeks
Population: All participants were included.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Minimal Acupuncture: Control Sham/Minimal Acupuncture: Control group will receive sham/minimal acupuncture with low level electrical stimulation. The sham intervention (also described as minimal intervention) will use superficial needle insertion at body locations not recognized as true acupoints. Patients will be explained that various acupuncture treatment protocols will be tested including "minimal acupuncture", therefore, the control group will not be aware of receiving sham acupuncture. These described acupuncture treatments are well accepted treat
- Standard Acupuncture Treatment: Standard acupuncture treatment: protocol will include 4 gates plus GV 20 to reduce anxiety and help with relaxation and to assess acupuncture naïve patient's response to needles during their first acupuncture encounter. Subsequent visits would include administration of curious meridian Chong Mo paired with Yang Ming. 4 Hz low level electrical stimulation will be applied.
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment
Number analyzed (Participants) | 10 | 11
score on a scale | -2.08 (0.68) | -2.91 (0.59)

2. Secondary Outcome: Tolerability of Acupuncture in Women With Interstitial Cystitis/Painful Bladder Syndrom
Description: The total number of acupuncture sessions stopped due to poor tolerability of acupuncture
Time Frame: 0 weeks, 6 weeks
Population: All participants were included.
Measure: Number; unit: total number of sessions
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment
Number analyzed (Participants) | 10 | 11
total number of sessions | 0 | 0

3. Secondary Outcome: Safety of Acupuncture in Women With Interstitial Cystitis/Painful Bladder Syndrome
Description: The total number of adverse events experienced by women receiving acupuncture
Time Frame: 0 weeks, 12 weeks
Population: All participants were included.
Measure: Number; unit: total number of adverse events
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment
Number analyzed (Participants) | 10 | 11
total number of adverse events | 0 | 0

4. Other Pre Specified Outcome: Change in Urinary Microbiome
Description: A change in the urinary microbiome may be detected for responders to acupuncture compared with nonresponders.
Time Frame: 0 weeks, 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: We followed the clinicaltrials.gov definition of adverse events, and documented any untoward or unfavorable medical occurrence in any participant
Arm/Group | Minimal Acupuncture | Standard Acupuncture Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02232282/Prot_SAP_000.pdf